CLINICAL TRIAL: NCT00984373
Title: Epidemiological Study to Describe Approaches in Diagnosis, Treatment and Social Functioning of Schizophrenic Patients in Bulgaria
Brief Title: Epidemiology of Schizophrenia in Bulgaria
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NBG-SER-2009/1
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia epidemiology; Schizophrenic patients' social and health characteristics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to provide accurate, reliable information on schizophrenia clinical management in order to detect unmet medical needs of this disease in terms of:

* Patient characteristics.
* Diagnostic and treatment approaches: initial and subsequent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia
* Above 18 years
* Signed Informed consent

Exclusion Criteria:

* Below 18 years
* Consent refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Bulgaria (7):
  - Research Site, Burgas
  - Research Site, Pazardzhik
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vidin